CLINICAL TRIAL: NCT06714097
Title: Application of Digital Twins' Technology in Patients Who Had a Stroke, with Moyamoya Disease and with Cerebral Amyloid Angiopathy (CAA) During the Secondary Prevention Phase: a Proof of Concept Using a Randomized Control Trial (Clinical Study 6, STRATIF-AI Project)
Acronym: SMART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: SMART
Record Dates: First submitted 2024-11-07; First posted 2024-12-03 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Stroke; Moyamoya Disease; Cerebral Amyloid Angiopathy
Keywords: stroke; secondary prevention; digital twin; Moyamoya Disease; Cerebral Amyloid Angiopathy
MeSH Terms: conditions — Stroke; Moyamoya Disease; Cerebral Amyloid Angiopathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard secondary prevention + digital twin (Experimental): Patients allocated to this arm will receive the standard secondary prevention and will also use the STRATIF-AI app, which will integrate digital twin (DT) technology to improve patient management during the secondary prevention phase and to assist patients in understanding key concepts, such as: "Why should I care about a certain risk factor (e.g. blood pressure), and how can my lifestyle impact that risk factor? In other words, they will use the app to understand their medical situation, and to set personal goals.
  Interventions: Device: AI
- Standard secondary prevention only (Active Comparator): Patients allocated to this arm will receive only standard secondary prevention, which includes typical treatments and monitoring protocols used for patients with stroke, Moyamoya disease, and CAA.
  Interventions: Other: healthy dialogue

INTERVENTIONS:
Device: AI — STRATIF-AI apps will be used as an integral part of the dialogue with patients during thesecondary prevention phase
  Arms: Standard secondary prevention + digital twin
Other: healthy dialogue — Patients allocated to arm 2 will receive only standard secondary prevention, which includes typical treatments and monitoring protocols used for patients with stroke, Moyamoya disease, and CAA
  Arms: Standard secondary prevention only

SUMMARY:
The goal of this clinical trial is to obtain initial feedback on the implementation of the STRATIF-AI platform and digital twin in the secondary prevention phase in patients with stroke, Moyamoya disease and Cerebral amyloid angiopathy, including adults of both sexes.

The main questions it aims to answer is: how is the patients' experience regarding the use of the STRATIF-AI platform? Researchers will compare Arm 1, who use the STRATIF-AI app in addition to standard secondary prevention, against Arm 2, who receive standard secondary prevention only, to collect feedback regarding the platform usability.

Participants in the Arm 1 will:

* Complete cognitive and psychological assessments at the time of the first visit and after six months
* Follow the indications received from the clinician for standard secondary prevention
* Use the STRATIF-AI app daily for health management
* Optionally, purchase wearable devices that connect to the app.
* Participate in interviews at the six-month mark to share their experiences with the app.

Patients in the Arm 2 will:

* Complete cognitive and psychological assessments at the time of the first visit and after six months
* Follow the indications received from the clinician for standard secondary prevention

DETAILED DESCRIPTION:
AIMS

Patients in secondary prevention with Moyamoya, CAA and stroke admitted to the Cerebrovascular Disease Unit of Carlo Besta Neurological Institute will be enrolled and randomized 1:1 in the following two arms:

* Arm 1 is the intervention group: patients allocated to this arm will receive the standard secondary prevention and will also use the STRATIF-AI app, which will integrate digital twin (DT) technology to improve patient management during the secondary prevention phase and to assist patients in understanding key concepts, such as: "Why should I care about a certain risk factor (e.g. blood pressure), and how can my lifestyle impact that risk factor? In other words, they will use the app to understand their medical situation, and to set personal goals.
* Arm 2 is the control group: patients allocated to this arm will receive only standard seconda prevention, which includes typical treatments and monitoring protocols used for patients with stroke, Moyamoya disease, and CAA.

Patients will be screened and enrolled upon admission to the Cerebrovascular Disease Unit. They will complete a set of clinical, cognitive, and psychological evaluation, performed at the time point of enrolment (T0) and at a 6-months follow-up (T1).

Only for the Arm 1, a brief explanation about the use of the app will add about 30 minutes to the initial visit. Afterward, patients can use the app at their discretion to assist in self-care. The app also offers the option to connect to wearable devices.

This study involves the collection of quantitative and qualitative data as follows:

1. Quantitative data:

   * Cognitive status will be evaluated with Montreal Cognitive Assessment (MOCA) test
   * General health and disability status will be evaluated with Patient Reported Outcome Measures: Short Form Health Survey 36 (SF-36), WHO Disability Assessment Schedule (WHO DAS 2.0),
   * Psychological status will be evaluated with Center for Epidemiologic Studies Depression Scales (CES-D), General Anxiety Disorder 7-Item (GAD-7), Fatigue Severity Scale, Impact of Event Scale Revised (IES-R).
   * Clinical functioning will be evaluated using the modified Rankin scale (mRS) and the Clinical Functioning Information Tool (ClinFIT).

   Moreover, we will collect clinical variables such as: TFNE (Transient Focal Neurological Episodes), headache, seizures, hypertension, diabetes mellitus, dyslipidemia, obstructive sleep apnea (OSA), ischemic heart disease, atrial fibrillation, smoke, weight, height, body Mass Index (BMI), sedentariness, current use of estrogens and progestins, hyperhomocysteinemia, previous head injury, previous neurosurgery, previous blood transfusion, comorbidities, current medical therapy.
   * Data related to the index event will be collected: symptomatic or asymptomatic patient; type of index event, date of index event, age of onset, mRS for symptomatic patients.
   * Socio-demographic data will be also collected (age, gender, birth date, age at the first visit, date of the visit, race, level of education).
2. Qualitative data Semi-structured interviews will be developed and perform at T1 to obtain feedback from the end users (patients and/or caregivers) of the DT to understand their user experience.

Qualitative analysis of user experiences will be the main focus. The NVivo software will be used to identify topics and perform advanced queries.

ELIGIBILITY:
Inclusion Criteria:

* People aged ≥ 18
* Clinical and neuroradiological diagnosis of stroke (TAC or MR); diagnosis of CAA based on Boston 2.0 criteria; diagnosis of Moyamoya disease based on diagnostic criteria 2021.
* MOCA total score ≥ 23
* modified Rankin Scale (mRS) ≤ 2
* First-time patients at the Besta Institute
* Ability to sign informed consent
* Possibility of performing a brain MRI

Exclusion Criteria:

* Patients with transient neurological deficits that resolve within an hour and normal brain imaging
* Patient under legal protection or deprived of liberty by judicial or administrative decision
* Patient whose follow-up will be impossible
* Contraindication to magnetic resonance imaging and/or Digital subtraction angiography (DSA)
* Pregnant patients
* Known or suspected drug or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Feedback from users | 12 months
  To get initial feedback on the patients' experience regarding the use of the STRATIF-AIplatform in the secondary prevention phase.

SECONDARY OUTCOMES:
feedback to developers | 12 months
  feedback to development team. This will be used as a starting point for future studiesand for conversations with other clinics, politicians, and policy maker.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Istituto Neurologico Carlo Besta, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Elkefi S, Asan O. Digital Twins for Managing Health Care Systems: Rapid Literature Review. J Med Internet Res. 2022 Aug 16;24(8):e37641. doi: 10.2196/37641. PMID 35972776
- [Background] Herrgardh T, Madai VI, Kelleher JD, Magnusson R, Gustafsson M, Milani L, Gennemark P, Cedersund G. Hybrid modelling for stroke care: Review and suggestions of new approaches for risk assessment and simulation of scenarios. Neuroimage Clin. 2021;31:102694. doi: 10.1016/j.nicl.2021.102694. Epub 2021 May 7. PMID 34000646
- [Background] Marwaa MN, Guidetti S, Ytterberg C, Kristensen HK. Using experience-based co-design to develop mobile/tablet applications to support a person-centred and empowering stroke rehabilitation. Res Involv Engagem. 2023 Aug 24;9(1):69. doi: 10.1186/s40900-023-00472-z. PMID 37620982
- [Background] Prust ML, Forman R, Ovbiagele B. Addressing disparities in the global epidemiology of stroke. Nat Rev Neurol. 2024 Apr;20(4):207-221. doi: 10.1038/s41582-023-00921-z. Epub 2024 Jan 16. PMID 38228908
- See also: Related Info — https://stratif-ai.eu/en